CLINICAL TRIAL: NCT06801691
Title: The Next Step Towards the Elimination of Iodine Deficiency and Preventable Iodine-related Disorders in Europe
Acronym: EUthyroid2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: EUthyroid (Other)
Collaborators: EU Horizon (Unknown); UK Research and Innovation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 101095643_2
Record Dates: First submitted 2025-01-07; First posted 2025-01-30 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-01

CONDITIONS: Iodine Deficiency
Keywords: Prevention; Iodine Deficiency; Intervention Study; Complex Intervention; Adaptation to context; Awareness; Iodine intake; Nutrition education

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Teaching programme on iodine (Experimental): Educational materials: Iodine Feedback Tool, lecture on the topic of iodine and health, booklet, exercises, group assignments and a webpage
  Interventions: Other: Experimental: Intervention group

INTERVENTIONS:
Other: Experimental: Intervention group — Educational materials: Iodine Feedback Tool, lecture on the topic of iodine and health, booklet, exercises, group assignments and a webpage This is a pre/post intervention with no control group.

SUMMARY:
In the EUthyroid2 intervention, measures are being developed and implemented in educational settings across the UK, Germany, Slovenia, the Republic of Cyprus, Bangladesh, and Pakistan to effectively raise awareness of the risks associated with iodine deficiency. Each participating country will employ three measurement points. The intervention will be tailored to the specific contextual characteristics of each implementation site. A process evaluation utilizing a convergent parallel mixed methods design will be conducted, involving surveys of students and teachers, as well as semi-structured interviews.

DETAILED DESCRIPTION:
Detailed Description:

BACKGROUND: Iodine deficiency (ID) is a leading risk factor for thyroid disorders and developmental impairments in offspring. It is recognized as one of the most preventable causes of mental impairment in children. The EUthyroid2 project aims to contribute to the prevention of ID and its associated symptoms and disease burden in adolescents across Europe and beyond.

AIM: This project seeks to develop and implement an educational intervention in various educational settings, effectively raising awareness of the risks associated with iodine deficiency.

METHODS: The intervention will be conducted in each participating country, with three clusters (secondary schools, high schools, and vocational schools) per country. The goal is to achieve a final sample of 4500 study participants in all countries combined, involving one baseline measurement and two follow-up assessments (2-4 weeks and 6-8 months post-intervention). Data will be collected at all measurement points, with variations in implementation accounted for due to differences between countries. To ensure the intervention's functionality and effectiveness, the project will consider recommendations for developing complex interventions, appropriate theoretical frameworks, and conduct a context analysis. Outcome measures will include a newly developed iodine awareness questionnaire (primary outcome) and an iodine-specific food frequency questionnaire. Additionally, socio-demographic characteristics will be measured. Descriptive analyses will be performed on all variables, with subgroup and country-specific analyses computed. A process evaluation will assess the implementation process using a convergent parallel mixed methods design, inviting teachers and students to participate in an online questionnaire. Semi-structured interviews will further enrich this evaluation.

CONCLUSION/OUTLOOK: The results of the EUthyroid2 project may assist health authorities across participating countries in implementing effective strategies to reduce iodine deficiency and its associated risks. Ultimately, this could lead to a sustainable decrease in the disease burden induced by iodine deficiency.

ELIGIBILITY:
Inclusion Criteria:

* sufficient language skills to understand the study information, informed consent

Exclusion Criteria:

* none

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4500 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in awareness | T1 (baseline) to T2 (2-4 weeks) and T3 (6-8 months) in students (13-17 years)
  1. Change in awareness of iodine and iodine deficiency: Difference in iodine awareness is measured by an iodine awareness questionnaire. The scoring ranges from 1 to 22 points with higher scores indicating a better outcome of awareness.

SECONDARY OUTCOMES:
Changes between teaching modalities | T1 (baseline) to T2 (2-4 weeks) and T3 (6-8 months)
  Differences in iodine awareness between students taught module A vs module A+B vs module A+C vs module A+B+C. Changes in iodine awareness are assessed by the iodine awareness questionnaire. The scoring ranges from 1 to 22 points with higher scores indicating a better outcome of awareness.
Changes in vocational schools, high- and secondary schools | T1 (baseline) to T2 (2-4 weeks) and T3 (6-8 months)
  Differences in iodine awareness between students in vocational schools vs high schools vs secondary schools. Changes in iodine awareness are assessed by the iodine awareness questionnaire. The scoring ranges from 1 to 22 points with higher scores indicating a better outcome of awareness.
Change between age groups and gender distinctions | T1 (baseline) to T2 (2-4 weeks) and T3 (6-8 months)
  Differences in iodine awareness between girls vs boys. Changes in iodine awareness are assessed by the iodine awareness questionnaire.
  Differences in iodine awareness between 13-year-olds vs 14-year-olds vs 15-year-olds vs 16-year-olds vs 17-year-olds. Changes in iodine awareness are assessed by the iodine awareness questionnaire. The scoring ranges from 1 to 22 points with higher scores indicating a better outcome of awareness.
  Gender and age will be self-reported in a socio-demographic questionnaire.
Change in iodine intake | T1 (baseline) to T2 (2-4 weeks) and T3 (6-8 months)
  Dietary iodine intake is assessed through a food frequency questionnaire (FFQ), covering five main categories (cow's milk, fish, eggs, supplements, and salt) and regional components in each country. Each category is scored based on frequency (portions per day, week, or month), and individual sources are analyzed for iodine intake. For example, taking supplements 5-7 times a week or consuming a combination of multiple sources of cow's milk, fish and eggs a week may suggest sufficient intake. Regional differences are also considered, as salt is an iodine source in countries like Pakistan and Bangladesh, but not in the UK or Norway. The number of iodine sources will be compared before and after the intervention within each country, with a higher number of sources indicating a higher iodine intake). The number will differ according to the number of sources in each country.

CONTACTS AND LOCATIONS:
Locations (6):
- Bangladesh University of Health, Dhaka, Bangladesh
- Cyprus University of Technology, Limassol, Cyprus
- University Medicine Greifswald, Greifswald, Germany
- Islamia College Peshawar, Peshawar, Khyber Pakhtunkhwa, Pakistan
- University Medical Centre Ljubljana, Ljubljana, Slovenia
- University of Surrey; Queen's University Belfast, Guildford, United Kingdom